CLINICAL TRIAL: NCT02673255
Title: Safety and Efficacy of Two Tetanus-Diphtheria Vaccines for a Donor Hyper Immunization Program
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biomat USA, Inc. (Industry)
Collaborators: Hammond Clinical Trial Consulting, LLC (Unknown); Axio Research. LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GB-0115
Record Dates: First submitted 2016-01-29; First posted 2016-02-03 (Estimated); Last update posted 2021-07-20 (Actual); Status verified 2019-12

CONDITIONS: Healthy
Keywords: Plasma; Plasma Donor; Plasma Donation; Tetanus; Td; Immunoglobulin; Hyper-immunization
MeSH Terms: conditions — Tetanus | interventions — Tetanus Toxoid; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sanofi Pasteur (Tenivac) (Experimental): Tetanus and Diphtheria (Td) Vaccine, Manufacturer: Sanofi Pasteur (Tenivac), Dose: 0.5 mL, Route: Intramuscular (IM) in the deltoid muscle, Frequency: Every 90 days, Duration: 5 doses, 1 year.
  Interventions: Biological: Tetanus and Diphtheria (Td) Vaccine
- MassBiologics (Experimental): Tetanus and Diphtheria (Td) Vaccine, Manufacturer: MassBiologics, Dose: 0.5 mL, Route: Intramuscular (IM) in the deltoid muscle, Frequency: Every 90 days, Duration: 5 doses, 1 year.
  Interventions: Biological: Tetanus and Diphtheria (Td) Vaccine

INTERVENTIONS:
Biological: Tetanus and Diphtheria (Td) Vaccine

SUMMARY:
Many plasma donation centers have Tetanus immunization programs that are implemented in order to collect plasma with high levels of tetanus antibodies. The immunization program requires participants to receive multiple tetanus vaccinations over a period of time with the goal of hyper-immunizing them to tetanus. Their antibody-rich plasma is then used to manufacture a tetanus immunoglobulin product which helps with the prophylaxis and treatment of tetanus disease.

The Tetanus vaccine previously used for these programs is no longer being manufactured. Therefore, we must evaluate the safety and efficacy of a different vaccine when used for this purpose. The only other FDA approved Tetanus vaccines currently available for adults in the US are combination vaccines that also immunize against Diphtheria and/or Pertussis.

In this study, the investigators will evaluate two vaccines that are combinations of Tetanus and Diphtheria (Td). Investigators will not evaluate any vaccines containing Pertussis antigen. The vaccines to be evaluated are manufactured by MassBiologics and Sanofi Pasteur (Tenivac).

The package insert for these vaccines indicates they should be administered to previously vaccinated people once every 10 years. However, this study will evaluate whether they are safe and effective for dosing every 90 days.

The investigators hypothesize that at least 25% of study subjects will have a positive response to at least one of the five planned doses. Each vaccine will be evaluated separately.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18* years of age at Visit 1.
2. Subject has met all suitability criteria that would allow donation as a Normal Source Plasma donor
3. Subject has not been immunized for tetanus within the prior three (3) months
4. Subject is not participating in any other immunization program
5. Subject possesses a pre-existing antibody for tetanus of at least 0.15 IU/mL

Exclusion Criteria:

1. Pregnant.
2. Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
3. Subject has a hypersensitivity to components in the vaccine (e.g., thimerosal, latex, etc.)
4. Subject has history of a severe reaction to any immunization
5. Subject has a history of Guillain-Barré Syndrome
6. Subject is unable to read and/or write due to illiteracy or a physical impairment.
7. The Investigator concludes that the anticipated vaccination site (deltoid area) is not suitable for adverse event assessment

   * Or legal adult according to local law. Participants in NE limited to individuals age 19-69 years due to age of majority laws in NE.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with a positive tetanus titer response following immunization | Through study completion, average 18 months.
  A "positive response" is defined as a 4-fold increase if the pre-vaccination titer was less than or equal to 2.7IU/mL or a 2-fold increase if the pre-vaccination titer was greater than 2.7IU/mL

SECONDARY OUTCOMES:
Number of participants experiencing vaccine-related adverse events | Through study completion, average 18 months.
  Number of related adverse events will be compared with prescribing information for the vaccine and with historic data on adverse event rates among Normal Source plasma donors and Hyper-Immunized plasma donors. Severity grading of vaccine-related adverse events is based on a modified version of FDA guidance dated September 2007 titled "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials."

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Rosa-Bray, MD, Principal Investigator — Biomat USA, Inc. (Sponsor)
Locations (4):
- United States (4):
  - Biomat Bellflower, Bellflower, California
  - Biomat Lincoln, Lincoln, Nebraska
  - Biomat Clarksville, Clarksville, Tennessee
  - Biomat Salt Lake City 1, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes